CLINICAL TRIAL: NCT03984500
Title: A Comprehensive Program to Increase Sickle Cell Trait Knowledge and Awareness Among Parents of Young Children Identified in Newborn Screening
Brief Title: A Program to Increase Sickle Cell Trait Knowledge Among Parent of Young Children Identified in Newborn Screening
Acronym: SCTaware
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Creary (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Susan Creary, Assistant Professor of Pediatrics, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00000122; 1R03HL146877-01 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-13 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Sickle Cell Trait
Keywords: Sickle Cell Trait; Education
MeSH Terms: conditions — Sickle Cell Trait | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Other): During phase 1 of this study parents who attend in person education sessions will be recruited to have their standard sessions video-taped, timed, and reviewed by the SCTaware Team. Subjects will complete before and after education questionnaires that will then be reviewed to see how much participants learned about SCT, how education was not clear and/or appropriate (too much medical jargon). The SCTaware education will then be created based on review of these videos and participants' survey responses.
  For phase 2 of the study, the same recruitment strategy will be utilized. Participants will receive SCTaware and complete before and after questionnaires for evaluation. Participants in this phase will also complete follow-up questionnaires at 1 and 6 months.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — SCTaware education (Phase II) will be compared to Ohio's current in-person SCT education (Phase I).

SUMMARY:
This is a study for parents of young children with Sickle Cell Trait (SCT) identified by newborn screening who are referred and present for in person SCT education at the Institution.

The study will determine the feasibility of implementing a SCT education program (SCTaware) that is appropriate for all parents, including those with low base knowledge and low health literacy and then test if results in high and sustained SCT knowledge.

DETAILED DESCRIPTION:
This is a single center, observational study to develop an education program for parents of young children diagnosed with Sickle Cell Trait. This will be accomplish by evaluating the current Ohio education in-person program, and assessing, through a set of questionnaires, how much participants are understanding about this diagnosis.

During phase I of the study, participants will be video-taped, and a set of questionnaires will be answer before and after education is given. This data will then be analyzed by the SCT Team in order to develop the Program.

During phase II of the study, population with the same criteria as phase I will be enrolled, however they will receive the revised "SCTaware" education. Pre and post education questionnaires will also be answered. In addition, participants during this phase will receive follow-up calls at 1 and 6 months to complete additional surveys.

In addition, the investigators will be using the Decisional Conflict Scale (DCS) to explore if parents experience decisional conflict about whether or not to obtain SCT testing and if SCTaware reduces this conflict

ELIGIBILITY:
Inclusion Criteria:

1. Adult biological parents of children <3 years old with Hemoglobin S-trait identified by NBS who present for SCT education at NCH.
2. English proficiency will be required

Exclusion Criteria:

1. Parents who self-report that they do not have functional verbal English (report that they are not proficient) or if they request an interpreter for the education session.
2. Parents who have previously attended an education session about an abnormal hemoglobinopathy trait
3. Parents who self-report that they have a child with SCD
4. Parents who self-report that they have SCD.
5. Parents who report that they or their partner is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing of a Sickle Cell Trait education Program: The time required to train a sickle cell trait educator and to deliver the revised sickle cell trait education will be measured | 2 years
  The time required to train a sickle cell trait educator and to deliver the revised sickle cell trait education will be measured. The program will be feasible if the time to train the educator and deliver the education can be completed within the context of the current sickle cell trait education program in Ohio.
Parental Sickle Cell Trait Knowledge | 2 years
  Parental Sickle Cell Trait Knowledge will be measured before the education, immediately after the education, and 6 months after the education is provided using the 8-question Sickle Cell Trait Knowledge Assessment Measure. Parents that score 75% correct on this measure or higher will be considered to have high knowledge. The proportion of those parents who have high knowledge prior to the education will be compared to the percentage of parents that have high knowledge 6-months after receiving the education.

SECONDARY OUTCOMES:
Percentage of Parents who receive on-site Sickle Cell Trait testing | 2 years
  On-site sickle cell trait testing will be available for all parents and will be ordered for all parents who accept this testing. The percentage of enrolled parents that accept and obtain on-site testing will be measured by the number of parents who accept this testing divided by the total number of parents who receive the education.
Decisional Conflict Scale | 2 years
  Parents will complete the 16 item validated decisional conflict scale survey before and after education to measure if parents' confidence or difficulty in making the decision whether or not to be tested for sickle cell trait improved with sickle cell trait education. These results are reported as a total score, with 5 sub-scores (uncertainty, informed, values clarity, support, and effective decision sub-scores). The total score and the sub-scores range from 0-100, with a score of 0 indicating no conflict/uncertainty and a score of 100 indicating extreme conflict/uncertainty.
Parental Anxiety | 2 years
  Parents will complete the state trait anxiety short from survey before and after receiving sickle cell trait education to measure if the education reduces parents' state anxiety about having a child with sickle cell trait.
Sickle Cell Trait Testing Cost | 2 years
  Parents will complete the sickle cell trait needs assessment survey that includes an item that asks participants if the cost of sickle cell testing impacted their decision whether or not to be tested for sickle cell trait.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Creary, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abrams MA, Zajo KN, Beeman CM, O'Brien SH, Chan PK, Shen Y, McCorkle B, Johnson L, Chisolm D, Barnard-Kirk T, Mahan JD, Christian-Rancy M, Creary SE. A Health Literate Approach to Address Health Disparities: a Virtual Program for Parents of Children with Sickle Cell Trait. J Commun Healthc. 2022;15(2):112-120. doi: 10.1080/17538068.2022.2026056. Epub 2022 Jan 19. PMID 36275941

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03984500/Prot_SAP_000.pdf